CLINICAL TRIAL: NCT05274451
Title: A Phase 1 Study to Assess the Safety and Efficacy of LYL797, ROR1-Targeting CAR T Cells, in Adults With Relapsed and/or Refractory Solid-Tumor Malignancies
Brief Title: A Study to Investigate LYL797 in Adults With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pipeline Reprioritization
Sponsor: Lyell Immunopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYL797-101
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer; TNBC - Triple-Negative Breast Cancer; Non-small Cell Lung Cancer; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Non-Small Cell Carcinoma of Lung, TNM Stage 4; Advanced Breast Cancer; Advanced Lung Carcinoma; NSCLC; NSCLC, Recurrent; NSCLC Stage IV; Relapsed Cancer; Relapse/Recurrence; Recurrent Breast Cancer; Recurrent NSCLC; Platinum-resistant Ovarian Cancer; Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Endometrial Cancer; Endometrioid Tumor; High Grade Serous Carcinoma; Ovarian Epithelial Cancer
Keywords: CAR T-cell therapy; CAR T; CAR T-cell; CAR-T; CAR-T cell therapy; CAR-T cell; ROR1; ROR1+; ROR1 positive; cell therapy; immunotherapy; relapsed; refractory; solid tumor; advanced; metastatic; breast cancer; lung cancer; triple negative breast cancer; non small cell lung cancer; ovarian cancer; endometrial cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Recurrence; Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, dose-escalation and -expansion study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental LYL797 (Experimental): ROR1-targeted CAR T cells
  Interventions: Biological: LYL797

INTERVENTIONS:
Biological: LYL797 — LYL797 is an autologous, genetically (Gen-R™) and epigenetically (Epi-R™) reprogrammed ROR1-targeted chimeric antigen receptor (CAR) T-cell therapy

SUMMARY:
This study will evaluate the safety and tolerability of LYL797, a ROR1-targeted CAR T-cell therapy, in patients with ROR1+ relapsed or refractory triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), platinum-resistant epithelial ovarian cancer/ fallopian tube cancer/ primary peritoneal cancer (Ovarian cancer), or Endometrial cancer. The first part of the study will determine the safe dose for the next part of the study, and will enroll patients with TNBC, NSCLC, Ovarian or Endometrial cancer. The second part of the study will test that dose in additional patients with TNBC, NSCLC, Ovarian or Endometrial cancer.

DETAILED DESCRIPTION:
This Phase 1, single-arm, open-label, multi-center, dose-escalation and expansion study will evaluate the safety and tolerability of LYL797, ROR1- targeted CAR T cells, in adults with relapsed and/or refractory ROR1+ triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), Ovarian cancer, or endometrial cancer. The dose-escalation phase includes patients with TNBC, NSCLC, Ovarian, or Endometrial cancer, and will investigate multiple dose levels to identify the recommended Phase 2 dose (RP2D). The dose-expansion phase will enroll patients with TNBC, NSCLC, Ovarian, or Endometrial cancer at the RP2D.

ELIGIBILITY:
IInclusion Criteria:

* ≥ 18 years of age at time of informed consent
* Confirmation of ROR1 expression from a pretreatment tumor sample
* Histologically confirmed TNBC or NSCLC that is relapsed or refractory, metastatic or locally advanced and unresectable
* Platinum-resistant epithelial ovarian cancer/ fallopian tube cancer/ primary peritoneal cancer.
* Endometrial cancer.
* Measurable disease including a target lesion and an additional lesion for biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ and marrow function
* Women of childbearing potential must have a negative pregnancy test at screening
* All participants must agree to practice highly effective methods of contraception

Exclusion Criteria:

* Prior treatment with any adoptive T-cell therapy or other anti-ROR1 therapy
* Prior solid organ transplantation
* Active, untreated brain metastasis or leptomeningeal disease; however, stable, treated brain metastases are allowed
* Untreated or active infection at the time of screening or leukapheresis
* HIV-positive, HTLV-1-positive, active acute HAV, acute or chronic HBV or HCV, or active tuberculosis
* Impaired cardiac function or clinically significant cardiac disease
* Uncontrolled pleural effusion, pericardial effusion, ascites requiring recurrent drainage procedures (once monthly or more frequent), or lymphangitis carcinomatosis
* History of interstitial pneumonitis or pulmonary fibrosis.
* Systemic corticosteroids or other immunosuppressive medications within 14 days of leukapheresis
* Pregnant or lactating/nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Evaluate incidence of dose-limiting toxicities (DLTs) | Up to 28 days
  Incidence of dose-limiting toxicities (DLTs)
Evaluate incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence of treatment-emergent adverse events (TEAEs)
Evaluate severity of treatment-emergent adverse events (TEAEs) | Up to 2 years
  Severity of treatment-emergent adverse events (TEAEs)
Determine recommended Phase 2 Dose (RP2D) | Up to 2 years
  Dose-escalation phase to determine the recommended Phase 2 dose

SECONDARY OUTCOMES:
Evaluate anti-tumor activity of LYL797 based on overall response rate (ORR) by RECIST, version 1.1 | Up to 2 years
  Overall response rate (ORR) by RECIST, version 1.1
Evaluate duration of response (DOR) | Up to 2 years
  Duration of response (DOR)
Evaluate progression-free survival (PFS) | Up to 2 years
  Progression-free survival (PFS)
Evaluate overall survival (OS) | Up to 2 years
  Overall Survival (OS)
Evaluate maximum concentration of LYL797 (Cmax) of LYL797 in peripheral blood (PB) samples | Up to 2 years
  Maximum concentration of LYL797 (Cmax)
Evaluate time to Cmax (Tmax) of LYL797 in peripheral blood (PB) samples | Up to 2 years
  Time to Cmax (Tmax)
Evaluate area under the concentration-time curve (AUC) of LYL797 in the peripheral blood (PB) | Up to 2 years
  Area under the concentration-time curve (AUC)
Evaluate Persistence of LYL797 CAR T cells in peripheral blood samples | Up to 2 years
  Time to last detectable LYL797, Tlast

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Walling, MBChB, PhD, Study Director — Lyell Immunopharma, Inc.
Locations (18):
- United States (18):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Los Angeles, Santa Monica, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Sidney Kimmel Cancer Center, Jefferson University Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute and Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No